CLINICAL TRIAL: NCT00541177
Title: Pilot Study of Prevention Myopia in Children With Low Concentration of Atropine
Brief Title: Study of Myopia Prevention in Children With Low Concentration of Atropine
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB960209-3
Record Dates: First submitted 2007-10-06; First posted 2007-10-10 (Estimated); Last update posted 2007-10-10 (Estimated); Status verified 2007-10

CONDITIONS: Myopia
Keywords: prevention myopia
MeSH Terms: conditions — Myopia | interventions — Atropine; Tropicamide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): use 0.25% atropine once a week
  Interventions: Drug: atropine
- 2 (Active Comparator): use 0.5% tropicamide everyday
  Interventions: Drug: tropicamide

INTERVENTIONS:
Drug: atropine — 0.25% atropine
  Arms: 1
Drug: tropicamide — 0.5% tropicamide
  Arms: 2

SUMMARY:
The purpose of this study is to test the hypothesis that myopia can be prevented by using a low concentration of atropine eyedrops once a week.

DETAILED DESCRIPTION:
The prevalence rate of myopia is rising rapidly in several Asian countries. A prevalence survey conducted in 1995 of 11178 school children in Taiwan were 12 percent for six year old and 84 percent for teenagers 16 o 18 years. Among them, twenty percent were high myopes. While in the United States and Europe the prevalence rate in older adults is 20% to 50%. The rate of progression of myopia is highest in young children, and the average age of stabilization of myopia is approximately 16 years.The onset of myopia may occur at a relatively young age, leading to higher risks of high myopia (myopia at least 6.0 diopters ) in adulthood. High myopia is associated with potentially blinding complications. Therefore, prevention of myopia progression is important in Taiwan, especially in young children.

There is some evidence that atropine eyedrops retard myopia progression in three randomized clinical trials. It is believed that atropine act on muscarinic receptor located in the sclera and through some unknown mechanism retard the elongation rate of axial length. However, the possible long-term side effects such as cataract formation and retinal toxicity, are largely unknown. Photophobia in daily life, accommodation difficulty both decrease the acceptance of atropine usage and compliance.

There are some evidence that the rate of axial elongation of eyeball are different between pre-myopic stage and myopic stage. Therefore, if we can use low concentration of atropine eyedrops before myopia development. Maybe we can prevent abnormal axial length elongation with lower dosage of atropine eyedrops compared with daily use of atropine eyedrops in true myopia stage.

Clinical study was conducted by randomized control trial. 60 school-aged children were recruited ( Age 7 to 12 years ). All with pre-myopia ( spherical equivalent between +0.50 and -0.75 ) after cycloplegic refraction. Visual acuity of naked eyes are above 0.6. None of them had tropia, amblyopia, eyelid disease, ocular problems. The astigmatism was less than -1.0D and anisometropia was less than 1.0D. The children were randomly assigned into two groups by using randomized consent design. The first group use 0.25% atropine once a week. The second group keep traditional treatment using 0.5% tropicamide eyedrop every day. All children had complete ophthalmologic examination before enrollment. Follow-up examinations were performed every 3 months for 12 months duration. These examinations included visual acuity of naked eye. Intraocular pressure, refractive status. The cycloplegic refraction and axial length were measured every 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Aged 7 to 12 years old
* Has pre-myopia (spherical equivalent between +0.50 and -0.75) after cycloplegic refraction.
* Visual acuity of naked eyes are above 0.6.
* Astigmatism is less than -1.0D and anisometropia less than 1.0D.

Exclusion Criteria:

* Has tropia, amblyopia, eyelid disease, or ocular problems.

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2007-04; Study Completion 2008-03 (Estimated)

PRIMARY OUTCOMES:
cycloplegic refraction, visual acuity | one year

SECONDARY OUTCOMES:
axial length | one year

CONTACTS AND LOCATIONS:
Overall Officials: Leon Chih-Kai Liang, MD MMS, Principal Investigator — Min-Sheng General Hospital; National Yang-Ming university, Taiwan
Locations (1):
- Min-Sheng General Hospital, Taoyuan District, Tao-Yuan, Taiwan